CLINICAL TRIAL: NCT02803164
Title: A Pilot Study to Evaluate the Efficacy of Vacuum-Assisted Dressings (V-AD) in the Management of Open Chest Wounds
Brief Title: Vacuum-Assisted Dressings (V-AD) in the Management of Open Chest Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mathew Thomas, M.D., PI, Mayo Clinic
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-002486
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Results first posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Open Chest Wounds
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Vacuum-assisted dressing (Other): Eligible subjects will receive negative pressure wound therapy during surgery.
  Interventions: Device: Wound Vacuum-assisted dressing
- Historical control group for comparison (Other): Retrospective review of subjects medical records with open chest wounds who were treated with the traditional treatment techniques.
  Interventions: Other: Control group

INTERVENTIONS:
Device: Wound Vacuum-assisted dressing — The NPWT system (V.A.C. Therapy System, KCI USA Inc.) consisted of a medical-grade non-adherent polyvinyl alcohol white foam applied directly to the infected surface, followed by an open-pore reticulated polyurethane black foam cut to fit the wound and covered by a transparent air-tight adhesive drape. A suction cup with tubing was placed over a small slit on the drape and connected to a suction machine (V.A.C. ULTA Therapy Unit).
  Other Names: Wound Vacuum-assisted dressing (V-AD)
  Arms: Vacuum-assisted dressing
Other: Control group — Retrospective review of subjects medical records with open chest wounds who were treated with the traditional treatment techniques.
  Arms: Historical control group for comparison

SUMMARY:
Vacuum-assisted dressings (V-AD) are effective in treating patients with open chest wounds (OCW) and will decrease the time-to-closure of such wounds when compared to a historical cohort of patients managed by traditional wound care management.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo surgical intervention(s) as part of the standard care for management of intra-thoracic infection.

Exclusion Criteria:

* Patent bronchopleural fistulas. Severe respiratory failure requiring mechanical ventilation at the time of first consultation.
* Proven or suspected malignancy in the wound. Coagulopathy due to medical or pharmacologic reasons. Dependency on anticoagulants or antiplatelet medication due to high risk for adverse events if these medications are stopped for a prolonged period of time.

Allergy to acrylic products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-11-03 (Actual); Study Completion 2020-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mauricia Buchanan, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Treatment of wound with Vacuum-assisted dressing.
  Wound Vacuum-assisted dressing: Management of chronic open chest wounds with V-AD assisted dressing.
- Historical Control: Retrospective review of subjects medical records with open chest wounds who were treated with the traditional treatment techniques
Period: Overall Study
Arm/Group | Intervention | Historical Control
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 21 completed
Groups:
- Control Group: Historical chest wound treatment.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control Group | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Median (Full Range); unit: years] | 61 [22 to 75] | 62 [18 to 77] | 62 [18 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 3 | 10 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Duration of Negative Pressure Wound Therapy (NWPT)
Description: The total number of days of receiving NWPT
Time Frame: 12 month follow up
Population: Data not collected or analyzed for the Historical Control arm. This arm did not receive the NWPT.
Measure: Median (Full Range); unit: Days
Arm/Group | Intervention | Historical Control
Number analyzed (Participants) | 10 | 0
Days | 8 [2 to 29] |

2. Secondary Outcome: Wound Closure
Description: The total number of days to wound closure
Time Frame: 12 months
Measure: Median (Full Range); unit: Days
Arm/Group | Intervention | Historical Control
Number analyzed (Participants) | 10 | 11
Days | 7 [4 to 49] | 18 [4 to 179]

3. Secondary Outcome: Length of Hospital Stay
Description: The total number of days in hospital
Time Frame: 12 months
Measure: Median (Full Range); unit: Days
Arm/Group | Vacuum-assisted Dressing | Historical Control Group for Comparison
Number analyzed (Participants) | 10 | 11
Days | 6 [1 to 43] | 25 [3 to 152]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention | Historical Control
All-Cause Mortality (participants affected / at risk) | 2/10 | 1/11
Serious Adverse Events (participants affected / at risk) | 2/10 | 11/11
Other Adverse Events (participants affected / at risk) | 2/10 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=10) | Historical Control (N=11)
Sepsis (Infections and infestations) | 1 (1) | 7 (7)
Major cardiac event (Cardiac disorders) | 0 (0) | 1 (1)
Air Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reintubation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute kidney failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=10) | Historical Control (N=11)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 5 (5)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Wound dehiscence (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT02803164/Prot_SAP_000.pdf